CLINICAL TRIAL: NCT04811846
Title: Circulating Tumor Cell (CTC) Quantification During Transurethral Resection (TURBT) and Plasma Kinetic Vaporisation (PKVBT) of Transitional Cell Carcinoma in Purging Fluid and Blood: a Randomized Controlled Trial
Brief Title: CTC Quantification During TURBT and PKVBT of Transitional Cell Carcinoma in Purging Fluid and Blood
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Teaching Hospital Hall in Tirol (Other)
Collaborators: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Gernot Ortner, Sub-Investigator, University Teaching Hospital Hall in Tirol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Urinary Bladder Neoplasm; Transitional Cell Carcinoma; Urogenital Neoplasms; Circulating Tumor Cell; Neoplasms
Keywords: Bladder cancer; NMIBC; CTC; Circulating tumor cell; Transurethral resection; Plasma kinetic vaporization; TURBT; PKVB
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Urogenital Neoplasms; Neoplastic Cells, Circulating; Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Pilot trial with parallel group design and comparison of 2 established techniques (TURBT, PKVB)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TURBT (Transurethral Resection of Bladder Tumor) (Active Comparator): For patients undergoing bipolar transurethral resection, bladder tumor is resected in a piecemeal manner.
  Interventions: Device: Bipolar transurethral resection of bladder tumor (TURBT)
- PKVB (Plasma Kinetic Vaporization of Bladder Tumor) (Active Comparator): For patients undergoing bipolar plasma kinetic vaporization of bladder tumor, bladder tumor is vaporized.
  Interventions: Device: Bipolar transurethral plasma kinetic vaporization of bladder tumor (PKVBT)

INTERVENTIONS:
Device: Bipolar transurethral resection of bladder tumor (TURBT) — Standard resection in piecemeal technique with standard bipolar cutting loop. (Storz medical, 27040 GP1)
  Arms: TURBT (Transurethral Resection of Bladder Tumor)
Device: Bipolar transurethral plasma kinetic vaporization of bladder tumor (PKVBT) — Vaporization of bladder tumor with standard bipolar vaporization electrode. (Storz medical, 27040 NB)
  Arms: PKVB (Plasma Kinetic Vaporization of Bladder Tumor)

SUMMARY:
Transurethral resection of bladder tumor (TURBT) is usually performed in a piecemeal technique. Tumor fragmentation and cell spilling could be responsible for high recurrence rates. Circulating tumor cells (CTCs) have been shown to be a prognostic predictor in disease progression in transitional cell carcinoma. In the current study the investigators aim to quantify CTCs in purging fluid and blood for recurrent intermediate risk bladder cancer during surgery for two different methods: TURBT and Plasma-kinetic vaporization of bladder tumor (PKVBT). Also correlations for recurrence will be investigated for the two different surgical methods.

DETAILED DESCRIPTION:
Bladder cancer is the 9th most commonly diagnosed cancer in men worldwide, with a standardized incidence rate of 9.0 per 100,000 person-years for men and 2.2 per 100,000 person-years for women. Amongst any caner entity, bladder cancer is the most expensive cancer regarding follow-up and life-time treatment costs due to the high probability of recurrence. Up to 85% of patients initially present with non muscle-invasive bladder cancer (NMIBC). Progression to muscle-invasive bladder cancer (MIBC) is up to 10-20%. NMIBC is characterized by a high risk of recurrence after transurethral resection of bladder tumor (TURBT): the 1-yr recurrence rate is 15-61% and the 5-yr recurrence rate is 31-78%. These numbers represent the heterogeneity of NMIBC.

Against any existing oncological principle, during TURBT bladder tumors are resected in a piecemeal manner. This results in tumor fragmentation and floating cancer cells inside the bladder during surgery. These cells may have the ability to re-attach on and re-implant into the bladder wall and may be responsible for early disease recurrence which is commonly seen after initial surgery. It has been shown that tumor cells may access the circulatory system through cut vessels. Circulating tumor cells (CTCs) can be detected in up to 20% in T1 high grade disease and are commonly seen in metastasized disease. They have shown to be an independent predictor of disease progression and relapse in several studies and reflect biological aggressiveness.

In the current study the investigators want to quantify CTCs for recurrent intermediate risk transitional cell carcinoma in purging fluid and blood for two different surgical methods: TURBT and Plasma-kinetic vaporisation of bladder tumors (PKVBT). Also correlations for recurrence will be investigated for the two different surgical methods.

In 2 urological centers (LKH Hall, LKH Salzburg) participants with diagnosed intermediate risk recurrent transitional cell carcinoma of the bladder will be randomly enrolled for either TURBT or PKVBT. Before surgery CTCs will be analyzed in peripheral blood and purging fluid. (preoperative CTCs blood and purging fluid, morphological aspect of CTCs in purging fluid) After resection for TURBT and vaporization for PKVBT, a tumor ground biopsy will be taken for both groups. After coagluation, CTCs will again be drawn in peripheral blood (intraoperative CTCs blood). After completion of surgery an indwelling catheter is inserted and purging fluid is again analyzed (postoperative CTCs purging fluid, morphological aspect of CTCs in purging fluid). Blood is again taken on day 2 after surgery during the morning routine to assess CTCs after surgery (postoperative CTCs blood). Patients will be dismissed on earliest day 2 after surgery after indwelling catheter removal.

Recurrence will be assessed during follow-up by cystoscopic controls (From 3 to 36 months after surgery). If recurrence is detected the study is terminated. If no recurrence is detected up to 36 months after surgery, the study is likewise terminated.

ELIGIBILITY:
Inclusion Criteria:

* female and male patients
* recurrent bladder tumor
* preoperative cystoscopy
* CT or MRI scan of abdomen not older than 30 days prior to surgery without suspicion of advanced disease (MIBC, metastasis)
* max. non-invasive papillary tumor (pTa) staging in prior histology
* max. low grade grading in prior histology
* max. 5 lesions in actual cystoscopy (all < 3cm)
* exophytic tumors
* transitional cell cancer of urinary bladder
* patient able to give consent
* signed consent form

Exclusion Criteria:

* initial tumor
* flat lesion
* > 3cm
* carcinoma in situ (CIS) in prior histology or suspicious CIS-finding in actual cystoscopy
* high grade grading in prior histology
* ≥ pT1 (tumor infiltration into subepithelial connective tissue) staging in prior histology
* > 5 lesions
* different entity from transitional cell carcinoma of urinary bladder
* prior radiation
* emergency surgery
* prior indwelling catheter (extraction < 1 week prior to surgery)
* pregnancy
* orthotopic neobladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-14 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
intraoperative CTC-number in blood [n/ml] | During surgery: after evacuation of snippets for TURBT and after full vaporization for PKVBT.
  Circulating tumor cells (CTCs) are measured in 15ml of peripheral blood which is taken during surgery. CTCs are quantified via automated immunofluorescence-microscopy. CK20+, p53+, DAPI+ and CD45- cells will be classified transitional cancer CTCs.
postoperative CTC-number in blood [n/ml] | 2nd postoperative day during morning routine.
  Circulating tumor cells (CTCs) are measured in 15ml peripheral blood which is taken after surgery. CTCs are quantified via automated immunofluorescence-microscopy. CK20+, p53+, DAPI+ and CD45- cells will be classified transitional cancer CTCs.
postoperative CTC-number in purging fluid [n/ml] | For both gruops (TURBT and PKVB) after insertion of indwelling catheter before finishing surgery.
  Circulating tumor cells (CTCs) are measured in purging fluid after the surgical intervention. After insertion of a new indwelling catheter the bladder is fully emptied and 100ml of sterile NaCl 0,9% is injected and extracted 5 times into and out of the bladder to mix CTCs. CTCs are quantified via automated immunofluorescence-microscopy. CK20+, p53+, DAPI+ and CD45- cells will be classified transitional cancer CTCs.
postoperative CTC morphology in purging fluid | After insertion of indwelling catheter before finishing the surgery.
  Cytological morphology of CTCs in purging fluid. CTCs will be examined for both groups and their morphological aspect (e.g. vital, non-vital, necrotic, deformed) is classified.
pre-to-intraoperative change of CTC-number in blood [n/ml] | Preoperative CTCs will be taken right before the start of surgery. Intraoperative CTCs will be taken after evacuation of snippets for TURBT and after full vaporization for PKVBT.
  The difference of the preoperative and intraoperative CTC-number in blood is calculated. Due to the intervention in both groups a difference in CTC-number is to be expected.
pre-to-postoperative change of CTC-number in blood [n/ml] | Preoperative CTCs will be taken right before the start of surgery. Postoperative CTCs will be taken on day 2 after surgery during the morning routine.
  The difference of the preoperative and postoperative CTC-number in blood is calculated. Due to the intervention in both groups a difference in CTC-number is to be expected.
intra-to-postoperative change of CTC-number in blood [n/ml] | Intraoperative CTCs will be taken after evacuation of snippets for TURBT and after full vaporization for PKVBT. Postoperative CTCs will be taken on day 2 after surgery during the morning routine.
  The difference of the intraoperative and postoperative CTC-number in blood is calculated. Due to the intervention in both groups a difference in CTC-number is to be expected.
pre-to-postoperative change of CTC-number in purging fluid [n/ml] | Preoperative CTCs in purging fluid are taken via an indwelling catheter right before start of the surgery. Postoperative CTCs in purging fluid are taken after insertion of a new indwelling catheter before finishing the surgery.
  The difference of the preoperative and postoperative CTC-number in purging fluid is calculated. Due to the intervention in both groups a difference in CTC-number is to be expected.

SECONDARY OUTCOMES:
Tumor recurrence [yes/no] | According to follow up cystoscopy at 3, 6, 12, 24, 36 months after intervention.
  Tumor recurrence is evaluated between 3 months and 36 months after surgery with follow-up cystoscopy.
Time to recurrence [days] | Through study completion, recurrence can occur within a maximum follow up of 36 months.
  The time difference from date of surgery to date of cystoscopic detection of recurrence. Including analysis of influencing factors.
preoperative CTC-number in purging fluid [n/ml] | Right before surgery.
  Circulating tumor cells (CTCs) are measured in purging fluid before the surgical intervention. After insertion of an indwelling catheter the bladder is fully emptied and 100ml of sterile NaCl 0,9% is injected and extracted 5 times into and out of the bladder to mix CTCs. CTCs are quantified via automated immunofluorescence-microscopy. CK20+, p53+, DAPI+ and CD45- cells will be classified transitional cancer CTCs.
preoperative CTC-number in blood [n/ml] | Right before start of surgery.
  Circulating tumor cells (CTCs) are measured in 15ml peripheral blood which is taken right before surgery. CTCs are quantified via automated immunofluorescence-microscopy. CK20+, p53+, DAPI+ and CD45- cells will be classified transitional cancer CTCs.
preoperative CTC morphology in purging fluid | Right before start of surgery.
  Cytological morphology of CTCs in purging fluid. CTCs will be examined for both groups and their morphological aspect (e.g. vital, non-vital, necrotic, deformed) is classified.

CONTACTS AND LOCATIONS:
Overall Officials: Udo Nagele, MD, Prof., Study Chair — Head of Department LKH Hall in Tirol; Lukas Lusuardi, MD, Prof., Study Chair — Heas of Department LKH Salzburg
Locations (2):
- Austria (2):
  - LKH Hall in Tirol, Department of Urology and Andrology, Hall in Tirol
  - LKH Salzburg, Department of Urology and Andrology, Salzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burger M, Catto JW, Dalbagni G, Grossman HB, Herr H, Karakiewicz P, Kassouf W, Kiemeney LA, La Vecchia C, Shariat S, Lotan Y. Epidemiology and risk factors of urothelial bladder cancer. Eur Urol. 2013 Feb;63(2):234-41. doi: 10.1016/j.eururo.2012.07.033. Epub 2012 Jul 25. PMID 22877502
- [Background] Comperat E, Larre S, Roupret M, Neuzillet Y, Pignot G, Quintens H, Houede N, Roy C, Durand X, Varinot J, Vordos D, Rouanne M, Bakhri MA, Bertrand P, Jeglinschi SC, Cussenot O, Soulie M, Pfister C. Clinicopathological characteristics of urothelial bladder cancer in patients less than 40 years old. Virchows Arch. 2015 May;466(5):589-94. doi: 10.1007/s00428-015-1739-2. Epub 2015 Feb 20. PMID 25697540
- [Background] Sylvester RJ, van der Meijden AP, Oosterlinck W, Witjes JA, Bouffioux C, Denis L, Newling DW, Kurth K. Predicting recurrence and progression in individual patients with stage Ta T1 bladder cancer using EORTC risk tables: a combined analysis of 2596 patients from seven EORTC trials. Eur Urol. 2006 Mar;49(3):466-5; discussion 475-7. doi: 10.1016/j.eururo.2005.12.031. Epub 2006 Jan 17. PMID 16442208
- [Background] Babjuk M, Bohle A, Burger M, Capoun O, Cohen D, Comperat EM, Hernandez V, Kaasinen E, Palou J, Roupret M, van Rhijn BWG, Shariat SF, Soukup V, Sylvester RJ, Zigeuner R. EAU Guidelines on Non-Muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol. 2017 Mar;71(3):447-461. doi: 10.1016/j.eururo.2016.05.041. Epub 2016 Jun 17. PMID 27324428
- [Background] Wilby D, Thomas K, Ray E, Chappell B, O'Brien T. Bladder cancer: new TUR techniques. World J Urol. 2009 Jun;27(3):309-12. doi: 10.1007/s00345-009-0398-9. Epub 2009 Mar 4. PMID 19259684
- [Background] Rink M, Schwarzenbach H, Vetterlein MW, Riethdorf S, Soave A. The current role of circulating biomarkers in non-muscle invasive bladder cancer. Transl Androl Urol. 2019 Feb;8(1):61-75. doi: 10.21037/tau.2018.11.05. PMID 30976570
- [Background] Engilbertsson H, Aaltonen KE, Bjornsson S, Kristmundsson T, Patschan O, Ryden L, Gudjonsson S. Transurethral bladder tumor resection can cause seeding of cancer cells into the bloodstream. J Urol. 2015 Jan;193(1):53-7. doi: 10.1016/j.juro.2014.06.083. Epub 2014 Jul 1. PMID 24996129
- [Background] Zare R, Grabe M, Hermann GG, Malmstrom PU. Can routine outpatient follow-up of patients with bladder cancer be improved? A multicenter prospective observational assessment of blue light flexible cystoscopy and fulguration. Res Rep Urol. 2018 Oct 9;10:151-157. doi: 10.2147/RRU.S141314. eCollection 2018. PMID 30349812
- [Background] Donat SM, North A, Dalbagni G, Herr HW. Efficacy of office fulguration for recurrent low grade papillary bladder tumors less than 0.5 cm. J Urol. 2004 Feb;171(2 Pt 1):636-9. doi: 10.1097/01.ju.0000103100.22951.5e. PMID 14713776
- [Background] Gazzaniga P, de Berardinis E, Raimondi C, Gradilone A, Busetto GM, De Falco E, Nicolazzo C, Giovannone R, Gentile V, Cortesi E, Pantel K. Circulating tumor cells detection has independent prognostic impact in high-risk non-muscle invasive bladder cancer. Int J Cancer. 2014 Oct 15;135(8):1978-82. doi: 10.1002/ijc.28830. Epub 2014 Mar 13. PMID 24599551
- [Background] Sievert KD, Amend B, Nagele U, Schilling D, Bedke J, Horstmann M, Hennenlotter J, Kruck S, Stenzl A. Economic aspects of bladder cancer: what are the benefits and costs? World J Urol. 2009 Jun;27(3):295-300. doi: 10.1007/s00345-009-0395-z. Epub 2009 Mar 7. PMID 19271220